CLINICAL TRIAL: NCT04719884
Title: Fluid Optimisation in Laparoscopic Colorectal Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Alenka Spindler-Vesel, asist prof, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 127/5/12
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Perioperative Complication
Keywords: postoperative complications, intraoperative monitoring, haemodynamic monitoring, laparoscopic abdominal surgery
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Standard perioperative anesthesia management
- Study group (Active Comparator): Perioperative extended haemodynamic monitoring of fluid loading, cardiac output and changes of peripheral vascular resistance by analysing the arterial curve was provided by non-invasive haemodynamic monitoring (LIDCO Rapid, Lidco Ltd., United Kingdom).In SG fluid optimisation was performed before pneumoperitoneum and after abdominal desuflation with actions to achieved CI, MAP and SI within 80% of baseline values.
  Interventions: Procedure: Perioperative fluid optimisation

INTERVENTIONS:
Procedure: Perioperative fluid optimisation — In case of stroke volume variation (SVV) >10% and SI and CI >10% below the starting value, fluid challenge was performed with approximately 2 ml/kg of colloid over maximum of 5 minutes. The response was monitored.
  If there was a fall in SVV and an increase in SI of >10% and the SVV still >10%, the second fluid challenge was performed.
  If there was still a reduction in SVV after the second fluid challenge, but an increase in nSI <10% and decrease in systemic vascular resistance (SVR), no additional fluids were given. Vasoactive drugs were used instead.
  Arms: Study group

SUMMARY:
Goal-directed fluid therapy (GDFT) with hemodynamic monitoring may not be of benefit to all elective patients undergoing major abdominal surgery, particularly those managed in Enhanced Recovery After Surgery protocols (ERAS) setting.

DETAILED DESCRIPTION:
Our study compared two groups of patients undergoing elective laparoscopic colorectal surgery: a control group (CG) in which standard haemodynamic monitoring was used, and a study group (SG) in which extended haemodynamic monitoring was applied with appropriate intraoperative interventions. Differences in intraoperative fluid management, hospital stay, and postoperative morbidity were observed.

ELIGIBILITY:
Inclusion Criteria:

* patients, undergoing elective laparoscopic colorectal surgery

Exclusion Criteria:

* Patients with cardiac arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Duration of hospitalisation | 1 month after admission

SECONDARY OUTCOMES:
Perioperative complications | 8 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Alenka Spindler Vesel, asoc Prof, Study Chair — Department of anesthesiology and surgical intensive care
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No